CLINICAL TRIAL: NCT01408004
Title: A Randomized Phase II Study to Explore the Efficacy and Feasibility of Upfront Bi-monthly Rotations Between Everolimus and Pazopanib in Patients With Advanced or Metastatic Clear Cell Renal Cancer
Brief Title: Rotating Pazopanib and Everolimus to Avoid Resistance
Acronym: ROPETAR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Netherlands Working Group on Immunotherapy of Oncology (Other)
Responsible Party: Principal Investigator, Prof. dr. E.E. Voest, Prof. dr. E.E. Voest, Netherlands Working Group on Immunotherapy of Oncology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL35303.041.11
Record Dates: First submitted 2011-04-07; First posted 2011-08-02 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Clear Cell Renal Carcinoma
Keywords: Renal carcinoma; Resistance; Reversible; Translational
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alternating regimen (Experimental): In the experimental arm (Arm A) alternating treatment will consist of 8 weeks of Pazopanib 800 mg qd alternated by 8 weeks of Everolimus 10 mg qd until first progression(PD per RECIST 1.1)followed thereafter by Pazopanib (when PD after 8 weeks of Everolimus)or Everolimus (when PD after 8 weeks of Pazopanib) monotherapy until second progression.
  Interventions: Drug: Pazopanib; Drug: Everolimus
- Sequential treatment (Active Comparator): The comparative arm (Arm B) will be the standard regimen of Pazopanib (800 mg qd continuously) until progression, followed thereafter by Everolimus (10 mg qd continuously) until progression.
  Interventions: Drug: Pazopanib; Drug: Everolimus

INTERVENTIONS:
Drug: Pazopanib — Tablet 800mg qd til progression
  Other Names: Votrient; L01XE11
  Arms: Sequential treatment
Drug: Everolimus — tablet 10 mg qd til progression
  Other Names: Afinitor; L01XE10
  Arms: Sequential treatment
Drug: Pazopanib — tablet 800mg qd, alternating schedule: 8 weeks Pazopanib, 8 weeks Everolimus
  Other Names: Votrient; L01XE11
  Arms: Alternating regimen
Drug: Everolimus — tablet 10mg qd, alternating schedule: 8 weeks Pazopanib, 8 weeks Everolimus
  Other Names: Afinitor; L01XE10
  Arms: Alternating regimen
Drug: Everolimus — Everolimus 10mg qd monotherapy until second progression (PD per RECIST 1.1)when first progression after 8 weeks of Pazopanib in alternating regimen
  Other Names: Afinitor; L01XE10
  Arms: Alternating regimen
Drug: Pazopanib — Pazopanib 800mg qd monotherapy until second progression (PD per RECIST 1.1) when first progression after 8 weeks of Everolimus in alternating regimen
  Other Names: Votrient; L01XE11
  Arms: Alternating regimen

SUMMARY:
In this study will be examined whether alternating treatment between two classes of drugs (TKI's and m-TOR inhibitors) postpones or prevents drug resistance in patients with renal cancer.

DETAILED DESCRIPTION:
Current practice is to treat with VEGFR-TKI or mTOR inhibitors until progression and then continue with the next active agent. From a biological perspective, TKI's will most likely activate compensatory pathways which, may ultimately lead to the development of resistance. Recent studies suggest that resistance to treatment with TKI may be reversible after stopping treatment. There is therefore a rationale to alternate treatment to prevent or delay the occurrence of resistance.

Our hypothesis is that alternating active agents in clear cell renal carcinoma (ccRCC) may reduce side effects, improve tolerability and compliance of treatment and prolong progression free survival and overall survival compared to the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up.
* Age ≥ 18 years.
* Histologically confirmed diagnosis of progressive metastatic clear cell renal cell cancer defined as >10% of the tumor cells having the clear cell phenotype.
* Locally advanced (defined as disease not amenable to curative surgery or radiation therapy) or metastatic RCC (equivalent to Stage IV RCC according to AJCC staging).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Measurable disease.
* No prior systemic anti-cancer treatment against clear cell renal carcinoma.
* Adequate organ system function.
* Non-childbearing potential.

Exclusion Criteria:

* Prior malignancy.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding.
* Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product.
* Presence of uncontrolled infection.
* Known past or present infection with Hepatitis B virus (HBV), Hepatitis C virus (HCV) or Human Immunodeficiency Virus (HIV).
* Corrected QT interval (QTc) > 480 msecs using Bazett's formula.
* History of one or more of the following cardiovascular conditions within the past 6 months:

  1. Cardiac angioplasty or stenting
  2. Myocardial infarction
  3. Stable or unstable angina pectoris.
  4. Coronary artery bypass graft surgery.
  5. Symptomatic peripheral vascular disease
  6. Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA).
* Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥160 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].
* History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.
* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any nonhealing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
* Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications or modify the dosing of interacting drugs for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Pregnant or lactating female.
* Treatment with any of the following anti-cancer therapies: Radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of Pazopanib OR Chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2011-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Randomization until earliest date of disease progression (according RECIST 1.1 criteria) or death, an expected average of one year

SECONDARY OUTCOMES:
Time to second progression | Time between first and second progression, an expected average of five months
  Time between first progression and second progression (PD) per RECIST 1.1 on Everolimus monotherapy (when PD after 8 weeks Pazopanib) or Pazopanib monotherapy (when PD after 8 weeks Everolimus) as second line treatment in experimental arm and time to progressive disease on Everolimus as second line treatment in comparative arm.
Change in Quality of life assessed by the FKSI-DRS and EORTC QLQ-C30 questionnaires compared to baseline | From randomization until one month after ceasing study medication, an expected average of 18 months
  Quality of life will be assessed bi-monthly by using the FACT Kidney Symptom Index (FKSI)-Disease Related Symptom (DRS)and the EORTC QLQ-C30 questionnaire. The symptoms covered by the FKSI-DRS include fatigue, pain, weight loss, dyspnea, cough, fever and hematuria. The EORTC QLQ-C30 questionnaire evaluates five functional scales (physical, role, emotional, social and cognitive functioning), three symptom scales (fatigue, pain, nausea, and vomiting), a global health status/QoL scale, and six single items (dyspnea, diarrhea, constipation, anorexia, insomnia and financial impact).
Toxicity reported as number/percentage of patients with adverse events | From randomization until one month after ceasing study medication, an expected average of 18 months
  Adverse events will be reported according Criteria for Adverse Events v4.0 (NCI CTCAE v4)
Overall survival | Time between randomization and death, an estimated average of 2-5 years

CONTACTS AND LOCATIONS:
Overall Officials: E.E. Voest, MD/PhD, Principal Investigator — UMC Utrecht
Locations (17):
- Netherlands (17):
  - St. Franciscus Gasthuis, Rotterdam, South Holland
  - UMC Utrecht, Utrecht, Utrecht
  - Medisch Centrum Alkmaar, Alkmaar
  - Acedemisch Medisch Centrum Amsterdam, Amsterdam
  - NKI-AVL, Amsterdam
  - Amphia ziekenhuis Breda, Breda
  - Maxima Medisch Centrum, Eindhoven
  - UMC Groningen, Groningen
  - Atrium Medisch Centrum Heerlen, Heerlen
  - Medische Centrum Leeuwarden, Leeuwarden
  - Acedemisch ziekenhuis Maastricht, Maastricht
  - St. Antonius ziekenhuis, Nieuwegein
  - Erasmus Medisch Centrum, Rotterdam
  - Orbis Medisch Centrum, Sittard-Geleen
  - Haga Ziekenhuis, The Hague
  - St. Elisabeth ziekenhuis, Tilburg
  - Isala klinieken, Zwolle

REFERENCES:
- [Derived] Cirkel GA, Hamberg P, Sleijfer S, Loosveld OJL, Dercksen MW, Los M, Polee MB, van den Berkmortel F, Aarts MJ, Beerepoot LV, Groenewegen G, Lolkema MP, Tascilar M, Portielje JEA, Peters FPJ, Klumpen HJ, van der Noort V, Haanen JBAG, Voest EE; Dutch WIN-O Consortium. Alternating Treatment With Pazopanib and Everolimus vs Continuous Pazopanib to Delay Disease Progression in Patients With Metastatic Clear Cell Renal Cell Cancer: The ROPETAR Randomized Clinical Trial. JAMA Oncol. 2017 Apr 1;3(4):501-508. doi: 10.1001/jamaoncol.2016.5202. PMID 27918762
- See also: Dutch Immunotherapy consortion for oncology — http://www.win-o.nl